CLINICAL TRIAL: NCT05902442
Title: A Clinical Comparison of Patient-specific 3D Printed Splints Versus Conventional Splints in the Treatment of Distal Radius Fractures.
Acronym: 3DxSPLINT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL83500.091.22
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Distal Radius Fractures
Keywords: 3D printing technology; Cast; Splint; Immobilization; Nonoperative; Patient specific; Radius Fracture
MeSH Terms: conditions — Wrist Fractures; Radius Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3DxSPLINT (Experimental)
  Interventions: Device: 3DxSPLINT

INTERVENTIONS:
Device: 3DxSPLINT — Routine immobilization procedure with a patient-specific 3D printed splint instead of the use of a conventional forearm splint after one week of conventional immobilization.

SUMMARY:
The goal of this clinical trial is to assess patient reported outcome measures of adult patients who are diagnosed with a distal radius fracture and treated with a patient-specific 3D printed splint as compared to a control cohort.

Patients receive routine immobilization procedure with a patient-specific 3D printed splint instead of the use of a conventional forearm splint after one week of conventional immobilization.

The main study parameters are patient reported outcome measures related to comfort and satisfaction of the medical aid. This will be measured qualitatively with a semi-structured interview and quantitively using questionnaires.

DETAILED DESCRIPTION:
Distal radius fracture (DRF) is a very common injury of the upper extremity. Yearly, over 45,000 patients visit the outpatient clinic with a DRF in the Netherlands. One third of these fractures are non-displaced and two thirds are displaced fractures. The conservative treatment of DRFs includes immobilization of the injured extremity using a conventional forearm cast. These casts do cause all sorts of discomfort during wear and impose life-style restrictions on the wearer. Examples are irritation and itching of the skin, pain from pressure points and inability to shower or swim without a protective sleeve. Emergent three-dimensional (3D) technology enables patient-specific splint design and fabrication. These splints are custom made to accurately fit the individual patient. The material of 3D printed splints is considered lightweight. Moreover, 3D splint design allows an open structure resulting in more ventilation, offering better hygiene and the possibility for wound control. The production of 3D splints can be accomplished with several hardware and software combination. The production process is similar overall and requires several steps. First image data with 3D spatial information of the limb is captured with either a 3D scanner or medical imaging device. The design of the 3D printed splint is further developed using a software application. The 3D splints design data is then exported, and the physical splint is printed using a 3D printer. Depending on material and device characteristics, postprocessing steps are required. The splint may require removal of support, curing and smoothing. If applicable, a closure mechanism is applied.

Currently most implementations of custom made 3D printed splints happen within the framework of case series or feasibility studies. Some previous studies have described on clinical tests from patients with promising results. However, studies are heterogenous in the use of hardware, software, 3D splint design, print materials, fabrication time and costs. Moreover, clinical comparison with conventional interventions remain scare. Therefore, it is challenging to determine the impact of 3D printed splints intervention on the patient with injuries .

The goal of this clinical trial is to assess patient reported outcome measures of adult patients who are diagnosed with a DRF and treated with a patient- specific 3D printed splint as compared to a control cohort. The secondary objectives are:

* To define whether treatment of 3D printed splints of DRF's result in the same clinical outcomes compared to treatment with standard plaster cast .
* To investigate the safety of 3D printed splint treatment.
* To generate hypothesis which individual characteristics might be used to determine which patients can benefit most from 3D printed splint treatment.
* To investigate barriers and facilitators to implementation.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years or older
* Admitted to the emergency department or plaster room with a DRF
* Non-operative treatment with cast immobilization
* Written informed consent
* Patients must be able to follow the study protocol

Exclusion Criteria:

* Operative treatment
* Open fractures
* History of surgically treated wrist fracture on the currently injured side within the last year (≤ 1 year)
* Unable to wear conventional forearm splint due to medical condition, known allergies or other reasons
* (partially) paralysis of the affected arm
* DRF older than two weeks

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
D-QUEST | three to five weeks post injury
  Instrument for measuring client satisfaction with a medical device. D-QUEST is a Dutch version of the Quebec User Evalutation of Satisfaction with assistive Technology.
CSD-OPUS | three to five weeks post injury
  The Orthotics and Prosthetics User's Survey on the Satisfaction with Devices.
EQ-5D VAS | three to five weeks post injury
  Rates the overall health of a patient.
Semi structured interview | three to five weeks post injury
  Patient reported outcome measrues related to comfort and satisfaction of the medical aid. Issures discussed:limitations daily life, cosmetic look and local complicaitons.

SECONDARY OUTCOMES:
PRWE | Approximately, one week, three to five weeks and 3 months post injury.
  Questionnaire to measure patient rated pain and disability for wrist conditions.
Complications | three months post injury.
  McKay checklist is used for scoring the complications after distal radius fracture.
Union rate | One week to three months post injury
  Union rate will be measured according to the current clinical standard.
Safety outcomes | one week to three months post injury
  Reasons for withdrawal and adverse events (production- and wearing of the 3D printed splints) are registered and evaluated
Barriers to implementation | one week to three months post injury
  Acceptance by caregivers and technical problems related to hardware- and software use in the 3D workflow are registered and evaluated.

OTHER OUTCOMES:
Baseline characteristics | Directly after admission
  Baseline characteristics as age, gender, fracture classification, side of fracture, dominant arm and activity of daily living are registerd.

CONTACTS AND LOCATIONS:
Overall Officials: V.M.A. Stirler, dr., Principal Investigator — Department of Trauma Surgery, Radboud University Medical Centre, Nijmegen, the Netherlands.

IPD SHARING:
Plan to Share IPD: Undecided